CLINICAL TRIAL: NCT04292574
Title: Spinal Muscular Atrophy Patient Registry of the United Kingdom and Ireland
Brief Title: UK SMA Patient Registry
Status: Recruiting | Type: Observational
Sponsor: Newcastle University (Other)
Collaborators: Biogen (Industry); Roche Pharma AG (Industry); Adult SMA REACH (Unknown); SMA REACH UK (Unknown)
Responsible Party: Sponsor
Other Study IDs: 22/NE/0131
Record Dates: First submitted 2020-02-28; First posted 2020-03-03 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Spinal Muscular Atrophy; SMA
Keywords: Spinal Muscular Atrophy; SMA; Neuromuscular Diseases; Motor Neuron Disease; Bulbo-Spinal Atrophy, X-Linked; Kennedy Disease; Spinal Muscular Atrophy with Respiratory Distress 1; Distal Spinal Muscular Atrophy; SMA type 1; SMA type 2; SMA type 3; SMA type 4; 5q SMA
MeSH Terms: conditions — Muscular Atrophy, Spinal; Neuromuscular Diseases; Motor Neuron Disease; Bulbo-Spinal Atrophy, X-Linked; Spinal muscular atrophy with respiratory distress 1; Spinal Muscular Atrophies of Childhood

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Spinal Muscular Atrophy
  Interventions: Other: Patient Registry

INTERVENTIONS:
Other: Patient Registry — Participants who have volunteered to participate will complete various questionnaires relating to their conditions.

SUMMARY:
Spinal muscular atrophy (SMA) is a form of motor neuron disease, most commonly caused by a mutation in the survival motor neuron 1 gene (SMN1) which results in a wide disease spectrum affecting children and adults. It is an autosomal recessive disorder and is therefore caused by inheritance of a mutated gene from each parent. All forms of SMA have an estimated combined incidence of 1 in 6,000 to 1 in 10,000 live births, with a carrier frequency of 1/40 to 1/60.

The patient registry aims to facilitate a questionnaire-based research study in order to better characterise and understand the disease in the UK and in Ireland. Entry is via self-registration over a secure internet connection (https://www.sma-registry.org.uk/). Online, patients are asked to read an information sheet about the research project and then indicate their consent to demonstrate willingness to participate. Following online consent, subjects will be entered into the registry. This is an on-going database and all participants are invited to update their information on a biannual basis.

DETAILED DESCRIPTION:
Participants are asked to provide information by completing online questionnaires. The medical questionnaire asks specific questions about their SMA diagnosis and their condition, including their motor function, requirement of assistance for feeding or breathing, scoliosis, contractures, hospitalisations, other illnesses, medications and participation in clinical trials. Additional short questionnaires collect information about patients' experience of daily life, their activities and quality of life, also known as patient-reported outcome measures or PROMs. Participants are asked to forward a copy of their genetic results to the registry.

The registry collaborates closely with the clinical networks SMA REACH UK (paediatric) and Adult SMA REACH and with TREAT-NMD Alliance.

The SMA REACH networks collect clinician-reported medical and functional assessment data from consented SMA patients who attend participating neuromuscular clinics in the UK. Links between the SMA REACH clinical databases and the UK SMA Patient Registry have been developed to enable the consented sharing of limited and specific data. Currently, linkage enables the sharing of patient-level PROMs data collected by the registry with each patient's SMA REACH clinic and with the SMA REACH coordination teams. At clinic level, the data informs patient care. At project coordination level, the data is aligned with clinical data collected by SMA REACH. It is then anonymised, analysed and reported to regulatory authorities as part of managed access agreements (MAA) for SMA therapies. Future linkage will enable patient registry participants to view elements of their own clinical data entered into the SMA REACH database by their doctor.

ELIGIBILITY:
Inclusion Criteria:

* All patients with a confirmed SMA diagnosis (or pending diagnosis) are eligible for inclusion. Diagnosis will be confirmed via genetic testing results

Exclusion Criteria:

* There are no exclusion criteria for the registry

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with SMA will volunteer to participate in this study. The study will be advertised through neuromuscular disease clinics, the registry website, patient organisations and conferences throughout the UK and Ireland.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2008-07-13 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Patient questionnaire | 12 months
  Patient-reported clinical and genetic confirmation of SMA, symptoms relating to muscle weakness, motor function, medication and family history. The patient registry collects the TREAT-NMD Expanded SMA Core Dataset, which includes post-marketing surveillance data items, and patient-reported outcome measures (PROMs).

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Marini-Bettolo, MD, PhD, Principal Investigator — Newcastle University
Locations (1):
- John Walton Muscular Dystrophy Research Centre, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Verhaart IEC, Robertson A, Wilson IJ, Aartsma-Rus A, Cameron S, Jones CC, Cook SF, Lochmuller H. Prevalence, incidence and carrier frequency of 5q-linked spinal muscular atrophy - a literature review. Orphanet J Rare Dis. 2017 Jul 4;12(1):124. doi: 10.1186/s13023-017-0671-8. PMID 28676062
- [Background] Verhaart IEC, Robertson A, Leary R, McMacken G, Konig K, Kirschner J, Jones CC, Cook SF, Lochmuller H. A multi-source approach to determine SMA incidence and research ready population. J Neurol. 2017 Jul;264(7):1465-1473. doi: 10.1007/s00415-017-8549-1. Epub 2017 Jun 20. PMID 28634652
- [Background] Muni-Lofra R, Murphy LB, Adcock K, Farrugia ME, Irwin J, Lilleker JB, McConville J, Merrison A, Parton M, Ryburn L, Scoto M, Marini-Bettolo C, Mayhew A. Real-World Data on Access to Standards of Care for People With Spinal Muscular Atrophy in the UK. Front Neurol. 2022 May 30;13:866243. doi: 10.3389/fneur.2022.866243. eCollection 2022. PMID 35707038
- See also: UK SMA Patient Registry website — https://www.sma-registry.org.uk/